CLINICAL TRIAL: NCT01660672
Title: A Dose-Escalation, Safety And Feasibility Study Of Enteral Levetiracetam For Seizure Control In Pediatric Cerebral Malaria
Brief Title: Enteral Levetiracetam For Seizure Control In Pediatric Cerebral Malaria
Acronym: LVT1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Gretchen Birbeck, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LVT1R01NS074409; 1R01NS074409-01A1 (NIH)
Record Dates: First submitted 2012-07-19; First posted 2012-08-09 (Estimated); Results first posted 2014-10-17 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-08

CONDITIONS: Seizure; Epilepsy; Cerebral Malaria
MeSH Terms: conditions — Seizures; Epilepsy; Malaria, Cerebral | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LEVETIRACETAM (Other): Open label, dose escalation to optimal dose.
  Interventions: Drug: LEVETIRACETAM

INTERVENTIONS:
Drug: LEVETIRACETAM — liquid, 40 mg/kg loading dose and 30mg/kg every 12 hours via nasogastric tube for 3 days--this is standard dose. If primary outcome is not reached, dose escalation to 150, 225, and 300% standard, as needed, will be conducted.
  Other Names: Keppra

SUMMARY:
Pediatric cerebral malaria (CM) affects more than 3 million children each year killing ~20% and leaving one third of survivors with long term neurologic and psychiatric sequelae. Seizures occur commonly with CM and are associated with an increased risk of death and neuropsychiatric disabilities. In this Malawi-based, dose- escalation, safety and feasibility study of enteral levetiracetam in pediatric CM, the investigators will lay the groundwork for future efficacy studies aimed at improving seizure control and ultimately decreasing the neurologic morbidity of pediatric CM.

DETAILED DESCRIPTION:
Cerebral malaria (CM) affects ~3 million children each year, primarily in sub-Saharan Africa. Antimalarial medications can rapidly clear P. falciparum parasites, but mortality rates remain high (12-25%). Survivors do not escape unscathed--~30% experience neurologic sequelae including epilepsy, behavioral disorders and gross neurologic deficits. Acute seizures occur commonly in CM and are associated with higher neurologic morbidity and mortality. Seizure management in malaria endemic regions is challenging because the available antiepileptic drugs (AED) induce respiratory suppression and assisted ventilation is unavailable. More optimal seizure control may improve neurologic outcomes in pediatric CM survivors, especially if the medication used is affordable and can be delivered safely and easily in resource limited settings. The investigators propose to conduct a dose- escalation, safety and feasibility study of enteral levetiracetam (LVT) for seizure control in children with CM and seizures admitted to Queen Elizabeth Central Hospital in Blantyre, Malawi. Enteral LVT given via nasogastric tube (NGT) rather than an intravenous (IV) formulation will be used since LVT has excellent enteral bioavailability and IV formations are not affordable in most malaria-endemic regions. LVT will be escalated based upon efficacy and toxicity endpoints with efficacy defined as seizure freedom in 75% of children during the 24 hours post LVT administration. Generally, only ~20% of children admitted with CM and seizures who receive standard AED treatment remain seizure free during the first 24 hours after admission. Safety assessments will include monitoring for problems related to NGT placement and medication delivery, laboratory parameters at 24 hours and 7 days post LVT, and overall case fatality rates. If efficacy endpoints are not met but enteral LVT is otherwise tolerated, LVT doses of ~3 times the standard dose used for other seizure-related conditions will be assessed. Pharmacokinetic (Pk) data on the absorption and elimination of LVT in CM will be obtained since enteral formulations are not typically used in critically ill children and malaria has been shown to impact drug absorption and elimination for some other medications. The safety, feasibility, Pk, optimal dosing and preliminary efficacy data from this proposed work will provide the information needed to determine whether to proceed with a randomized clinical trial of LVT in pediatric CM patients which would include acute seizure control as well as long term neurologic outcomes as critical endpoints. Since enteral LVT is relatively affordable for short-term use and could be feasibly delivered in resource limited settings, this therapy could potentially be scaled up for broad use throughout malaria endemic African countries

ELIGIBILITY:
Inclusion Criteria:

* Comatose with Blantyre Comas Score ≤ 3
* P. falciparum parasitemia
* Active seizure

Exclusion Criteria:

* Serum creatinine > 2mg/dL
* Pre-admission/concomitant treatment with antiretroviral medications for HIV (ARVs), antituberculous treatments(ATTs), or chronic use of any other enzyme-inducing medications

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen L Birbeck, M.D., Principal Investigator — University of Rochester
Locations (1):
- Queen Elizabeth Central Hospital, Blantyre, Malawi

REFERENCES:
- [Derived] Birbeck GL, Herman ST, Capparelli EV, Dzinjalamala FK, Abdel Baki SG, Mallewa M, Toto NM, Postels DG, Gardiner JC, Taylor TE, Seydel KB. A clinical trial of enteral Levetiracetam for acute seizures in pediatric cerebral malaria. BMC Pediatr. 2019 Nov 1;19(1):399. doi: 10.1186/s12887-019-1766-2. PMID 31672143

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LEVETIRACETAM
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LEVETIRACETAM
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: months] | 40.8 [27 to 71]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Region of Enrollment [Number; unit: participants]
  Malawi | 7

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Seizure
Description: Number of subjects free of seizure at 24 hours after initiation of treatment
Time Frame: 24 hours
Measure: Number; unit: individuals
Groups:
- LEVETIRACETAM: Open label, dose escalation to optimal dose.
  LEVETIRACETAM: liquid, 40 mg/kg loading dose and 30mg/kg every 12 hours via nasogastric tube for 3 days--this is standard dose.
Arm/Group | LEVETIRACETAM
Number analyzed (Participants) | 7
individuals | 7

2. Secondary Outcome: Toxicity Related to LVT
Description: Toxicity including vomiting, aspiration, complications related to the NGT, laboratory parameters at 24 hours and 1 week post LVT administration, and an overall acute case fatality rate significantly above the consistent historical ward average for CM. Pk studies to evaluate LVT absorption and elimination in pediatric CM.
Time Frame: 1 week
Measure: Number; unit: participants
Arm/Group | LEVETIRACETAM
Number analyzed (Participants) | 7
participants | 0

3. Secondary Outcome: Range of Plasma Concentration of LVT Across All Individuals
Description: Range of plasma LVT concentrations will be determined through HPLC method at eight timepoints post administration to evaluate LVT absorption and elimination in pediatric CM.
Time Frame: 72 hours
Measure: Mean (Full Range); unit: mcg/ml
Arm/Group | LEVETIRACETAM
Number analyzed (Participants) | 7
mcg/ml | 35 [20 to 50]

4. Other Pre Specified Outcome: Number of Participants With Neurologic Sequelae at Discharge
Description: Number of participants with neurologic sequelae at discharge
Time Frame: day 7
Measure: Number; unit: participants
Arm/Group | LEVETIRACETAM
Number analyzed (Participants) | 7
participants | 2

5. Other Pre Specified Outcome: Number of Subjects With Retinopathy at Enrollment
Description: Retinopathy status may impact LVT efficacy and subject status will be analyzed based on this characteristic.
Time Frame: Upon admission
Measure: Number; unit: participants
Arm/Group | LEVETIRACETAM
Number analyzed (Participants) | 7
participants | 4

6. Other Pre Specified Outcome: Number of Subjects Exposed to Phenobarbitone Prior to Enrollment
Description: Pre-enrollment exposure to phenobarbitone may impact LVT efficacy, and analysis base on this characteristic will be evaluated.
Time Frame: 0 hour
Measure: Number; unit: participants
Arm/Group | LEVETIRACETAM
Number analyzed (Participants) | 7
participants | 3

7. Other Pre Specified Outcome: Number of Participants Requiring AED During Admission
Description: Number of participants who required AEDS during admission(including for breakthrough seizures in the LVT group) during admission.
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | LEVETIRACETAM
Number analyzed (Participants) | 7
participants | 6

8. Other Pre Specified Outcome: Mean Time to Return to a BCS Score Greater Than or Equal to 4
Description: Mean time from admission to a BCS score greater than or equal to 4. The BCS (Blantyre Coma Scale) is a 0-5 scale measuring motor response, verbal response and eye movement assessing the severity of coma in children with cerebral malaria. Lower scores correspond to more profound coma.
Time Frame: 7 days
Measure: Mean (Full Range); unit: hours
Arm/Group | LEVETIRACETAM
Number analyzed (Participants) | 7
hours | 35.3 [7 to 78]

ADVERSE EVENTS:
Groups:
- LEVETIRACETAM: Open label, dose escalation to optimal dose.
  LEVETIRACETAM: liquid, 40 mg/kg loading dose and 30mg/kg every 12 hours via nasogastric tube for 3 days--this is standard dose. This dose was effective in 7/7 children.
Arm/Group | LEVETIRACETAM
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEVETIRACETAM (N=7)
Electrolyte (Blood and lymphatic system disorders) | 2 (3)
GI Symptoms (Gastrointestinal disorders) | 6 (6)
Hematologic abnormality (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No